CLINICAL TRIAL: NCT05174585
Title: A Phase 1/2a, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of Antitumor Activity of JAB-BX102 Monotherapy and Combination With Pembrolizumab in Adult Patients With Advanced Solid Tumors
Brief Title: JAB-BX102 Monotherapy and Combination With Pembrolizumab in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jacobio Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAB-BX102-1001; MK-3475-E58 (Other: Merck Sharp & Dohme LLC); KEYNOTE-E58 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor
Keywords: Solid Tumor; Anti-CD73 Monoclonal Antibody; CD73
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A, JAB-BX102 monotherapy, Phase 1, Dose Escalation (Experimental): Dose escalation of JAB-BX102 will be administered as monotherapy to determine the MTD and RP2D.
  Interventions: Biological: JAB-BX102 (anti-CD73 monoclonal antibody)
- Arm B, JAB-BX102 combination with pembrolizumab, Phase 2a, Dose Expansion (Experimental): JAB-BX102 will be administered in combination with pembrolizumab in specific solid tumor patients to evaluate the preliminary antitumor activity.
  Interventions: Biological: JAB-BX102 (anti-CD73 monoclonal antibody); Biological: pembrolizumab (anti-PD-1 monoclonal antibody)

INTERVENTIONS:
Biological: JAB-BX102 (anti-CD73 monoclonal antibody) — Administered by intravenous infusion (IV)
Biological: pembrolizumab (anti-PD-1 monoclonal antibody) — Administered by intravenous infusion (IV)
  Other Names: KEYTRUDA®
  Arms: Arm B, JAB-BX102 combination with pembrolizumab, Phase 2a, Dose Expansion

SUMMARY:
This study is to evaluate the safety and tolerability of JAB-BX102 monotherapy and combination therapy with pembrolizumab in adult participants with advanced solid tumors.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of JAB-BX102 monotherapy to determine the MTD(maximum tolerated dose) and RP2D(Recommended Phase 2 Dose) during Dose Escalation phase; then to evaluate preliminary antitumor activity when JAB-BX102 is administered in combination with pembrolizumab during Dose Expansion phase in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide an archived tumor sample
* Must have histologically or cytologically confirmed metastatic or locally advanced solid tumor
* Must be refractory to or become intolerant of existing therapy(ies) known to provide clinical benefit for their condition, or patient has no access to SOC treatment.
* Must have at least 1 measurable lesion per RECIST v1.1
* Must have adequate organ functions

Exclusion Criteria:

* Has central nervous system(CNS) metastases or carcinomatous meningitis, except if CNS metastases treated and no evidence of radiographic progression or hemorrhage for at least 28 days
* Active infection requiring systemic treatment within 7 days
* Active hepatitis C virus(HBV), hepatitis C virus(HCV), or HIV
* Any severe and/or uncontrolled medical conditions
* Left ventricular ejection fraction(LVEF) ≤50% assessed by echocardiogram (ECHO) or multigated acquisition scan (MUGA)
* QTcF(Corrected QT interval - Fredericia formula) interval >470 msec
* Experiencing unresolved CTCAE 5.0 Grade >1 toxicities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Dose Escalation phase Number of participants with dose limiting toxicities (DLTs) | First 21 days of Cycle 1
  A DLT is defined as the clinically significant TRAE(treatment-related adverse events) or abnormal laboratory values assessment during the first 21 days of Cycle 1 and excludes events that are deemed clearly related to underlying disease, progression, or intercurrent illness.
Dose Escalation and Dose Expansion phase: Number of participants with adverse events | Up to 3 years
  Patients will be assessed for incidence and severity of adverse events (AEs) according to NCI-CTCAE 5.0.
Dose Expansion phase: Overall response rate (ORR) | Up to 3 years - from baseline to RECIST confirmed Progressive Disease
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) per RECIST v 1.1.
Expansion phase: Duration of response (DOR) | Up to 3 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to disease progression per CTCAE v1.1 or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
To characterize the pharmacokinetics(PK) profile of JAB-BX102 as a single agent and in combination with pembrolizumab | Up to 3 years
  observed plasma concentration of JAB-BX102
Dose Escalation phase: Overall response rate (ORR) | Up to 3 years - from baseline to RECIST confirmed Progressive Disease
  The percentage of participants with complete response (CR) or partial response (PR) on RECIST v 1.1.
Dose Escalation phase: Duration of response (DOR) | Up to 3 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to disease progression per CTCAE v1.1 or death due to any cause, whichever occurs first.
Dose Escalation and Dose Expansion phase: Disease Control Rate (DCR) | Up to 3 years
  DCR is defined as percentage of participants with complete response (CR), partial response (PR), or stable disease (SD) per CTCAE v1.1.
Dose Escalation and Dose Expansion phase: Progression-free survival (PFS) | Up to 3 years
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression per CTCAE v1.1 or death which occurs first

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Huashan Hospital, Shanghai, Shanghai Municipality